CLINICAL TRIAL: NCT06438354
Title: Non-surgical Treatment of Residual Periodontal Pockets Using Sodium Hypochlorite/Amino Acid Gel and Cross-linked Hyaluronic Acid - a 9-month Randomized Controlled Clinical Trial.
Brief Title: Non-surgical Step 3 Periodontal Treatment With/Without Adjunctive Protocol - Pilot RCT.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Witten/Herdecke (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 64/2022
Record Dates: First submitted 2024-05-27; First posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Periodontal Pocket
MeSH Terms: conditions — Periodontal Pocket

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Test arm, patients undergo subgingival instrumentation of residual active site together with an adjunctive treatment protocol.
  Interventions: Biological: subgingival instrumentation plus Perisolv / hyaDent BG
- Group B (Placebo Comparator): Control arm, patients undergo subgingival instrumentation of residual active site only.
  Interventions: Procedure: subgingival instrumentation

INTERVENTIONS:
Biological: subgingival instrumentation plus Perisolv / hyaDent BG — Group A: Perisolv is applied prior to subgingival instrumentation for disinfecting purpose, hyaDent BG seals the site for accelerated blood clot stabilisation and support of cell proliferation.
  Arms: Group A
Procedure: subgingival instrumentation — Group B: sites requiring re-treatment are subjected to subgingival scaling
  Arms: Group B

SUMMARY:
Study conducted in patients recruited at private praxis setting after completed step 2 periodontal therapy. Residual pockets ≥4mm with positive bleeding or such >5mm randomly allocated to either conventional subgingival re-instrumentation (controls) or to same mechanical treatment with adjectively applied hypochlorite/aminoacid gel for antiseptic reason followed by subginigival placement of cross linked hyaluronic acid gel for sealing the site after instrumentation. Re-evaluations at 3 and 9 months controlled for clinical parameters such as Periodontal Probing Depth (PPD) (CAL), Clinical Attachment Level, Gingival Recession (GR), Bleeding on Probing (BOP). The hypothesis is, sites treated with adjunctive protocol show greater PPD reduction and greater CAL gain at 9-month evaluation.

ELIGIBILITY:
Inclusion Criteria:

* systemically healthy individuals, smokers and non-smokers, HbA1c <7.5%, compliant and adhering to systematic periodontal treatment protocol incl. SPT visits, patients willing to complete a 9-month post-op observation period

Exclusion Criteria:

* rheumatoid arthritis, HbA1c ≥7.5%, treatment of periodontitis within past 12 months, use of systemic antibiotics in past 6 months, pregnant and lactating individuals

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Clinical Attachment Level | 9 month post-op
  Greater amount of CAL gain in the test group A vs. control group B anticipated

SECONDARY OUTCOMES:
Periodontal Probing Depth | 9 months post-op
  Greater reduction in PPD for group A vs. Group B anticipated
Gingival Recession | 9 months post-op
  Similar change in the GR depth anticipated for both groups
Bleeding on Probing | 9 months post-op
  greater reduction in BOP anticipated for group A vs. group B patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Implantat Competence Centrum München, Munich, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ramanauskaite E, Machiulskiene V, Shirakata Y, Dvyliene UM, Nedzelskiene I, Sculean A. Clinical evaluation of sodium hypochlorite/amino acids and cross-linked hyaluronic acid adjunctive to non-surgical periodontal treatment: a randomized controlled clinical trial. Clin Oral Investig. 2023 Nov;27(11):6645-6656. doi: 10.1007/s00784-023-05271-0. Epub 2023 Sep 23. PMID 37740107
- [Result] Shirakata Y, Nakamura T, Setoguchi F, Imafuji T, Shinohara Y, Matsumura S, Iwata M, Noguchi K, Ramanauskaite E, Sculean A. Histological evaluation of nonsurgical periodontal treatment with and without the use of sodium hypochlorite / amino acids and cross-linked hyaluronic acid gels in dogs. Clin Oral Investig. 2024 Apr 27;28(5):281. doi: 10.1007/s00784-024-05674-7. PMID 38676852
- [Derived] Benyei L, Friedmann A, Ostermann T, Diehl D. Non-surgical treatment of residual periodontal pockets using sodium hypochlorite/amino acid gel and cross-linked hyaluronic acid-a 9-month pilot randomized controlled clinical trial. Clin Oral Investig. 2024 Sep 5;28(9):513. doi: 10.1007/s00784-024-05906-w. PMID 39235513